CLINICAL TRIAL: NCT05030389
Title: Effects of Long-term Remote Health Monitoring Through Bright Light Exposure, Physical Adapted Activity and Galvanic Vestibular Stimulation on the Sleep of the Elderly: Study Protocol for a Randomised Controlled Trial
Brief Title: Vestibular Stimulation, Exercise and Light Optimization for Circadian Clock Enhancement (Velocce)
Acronym: velocce
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Université de Caen Normandie (Other)
Collaborators: Région Normandie (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Université de Caen Normandie
Record Dates: First submitted 2021-06-25; First posted 2021-09-01 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-07

CONDITIONS: Healthy Aging
Keywords: Exercise; Biological rhythms; Vestibular stimulation
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Adapted Physical Activity (APA) (Experimental): Participants receive a web-based adapted physical activity (APA) during 12 weeks, on the basis of three at-home sessions a week
  Interventions: Behavioral: Adapted Physical Activity (APA)
- Adapted Physical Activity + Bright Light Exposure (APA + BLE) (Experimental): Participants receive a web-based APA program during 12 weeks on the basis of three at-home sessions a week, supplemented by a bright light exposure (BLE) during 12 weeks, on the basis of five at-home sessions a week
  Interventions: Behavioral: Adapted Physical Activity (APA); Behavioral: Bright Light Exposure (BLE)
- Galvanic Vestibular Stimulation (GVS) (Experimental): Participants receive Galvanic Vestibular Stimulation (GVS) during two weeks, on the basis of five at-home sessions a week
  Interventions: Behavioral: Galvanic Vestibular Stimulation (GVS)
- Health Education program (HE) (Active Comparator): Participants receive a web-based health education program (HE) during 14 weeks, on the basis of one at-home session a week
  Interventions: Behavioral: Health Education program (HE)

INTERVENTIONS:
Behavioral: Adapted Physical Activity (APA) — The APA program lasts 12 weeks and consists in three one-hour at-home sessions a week (total of 36 sessions), including two aerobic dominant web-based sessions and one muscle strengthening self-guided session.
  Arms: Adapted Physical Activity (APA); Adapted Physical Activity + Bright Light Exposure (APA + BLE)
Behavioral: Bright Light Exposure (BLE) — Bright light exposure (BLE) consists in using lamps for light therapy during 12 weeks, at the rate of five one-hour at-home sessions a week.
  Arms: Adapted Physical Activity + Bright Light Exposure (APA + BLE)
Behavioral: Galvanic Vestibular Stimulation (GVS) — The GVS program lasts 2 weeks and consists in five 20-minutes at-home sessions a week (total of 10 sessions), using a portable galvanic stimulator.
  Arms: Galvanic Vestibular Stimulation (GVS)
Behavioral: Health Education program (HE) — The HE program lasts 14 weeks and consists in one one-hour at-home session a week (total of 14 sessions). This web-based intervention includes courses on general health (sleep habits, diet, physical activity, cardiovascular diseases, etc.).
  Arms: Health Education program (HE)

SUMMARY:
This study investigates the effects of remote interventions based on the exposure to one or more zeitgebers (i.e. adapted physical activity alone or combined with bright light exposure, or galvanic vestibular stimulation) performed several times a week during three months on older adults' sleep and quality of life.

DETAILED DESCRIPTION:
More precisely, the main objective is to investigate the effects of interventions on objective sleep measures of older adults with a sleep complaint.

The main hypothesis is that the quantity and quality of sleep will be improved after the interventions in comparison to the active control group.

The second objective is to study the effects of these interventions on quality of life, physical condition, anxiety, depression and cognition.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer (men or women)
* Aged from 60 to 70 years
* Retired for at least 12 months
* Having a sleep complaint (overall score on the Pittsburgh Sleep Quality Index (PSQI) > 5, enquire information when these complaints appeared)
* Able to receive enlightened information in French and express consent
* Having a circadian typology of the "intermediate", "moderate morning" or "moderate evening" type, according to the circadian typology questionnaire of Horne and Ostberg (1976)
* Having cognitive abilities to understand oral instructions, objective by a Mini Mental State Examination (MMSE) score greater than or equal to 24
* Having a personal computer with a web cam, a microphone and an internet connection
* Living in Normandy
* Affiliated to the social security system
* French-speaking

Exclusion Criteria:

* Illiteracy
* Age-related macular degenerescence (AMD), blindness, visual acuity < 2 and other pathologies reducing the perception of light
* Bradycardia treatments (beta-blockers, digitalis, antiarrhythmics, bradycardic calcium channel blockers, etc.)
* Declaration of dementia (Alzheimer's disease, vascular dementia)
* Declaration of vestibular or neurological anomalies
* Declaration of progressive neurological disease (brain tumour, epilepsy, migraine, stroke, sclerosis, myoclonus, chorea, neuropathy, muscular dystrophies, myotonic dystrophy, Parkinson's disease)
* Declaration of pathologies with short-term vital prognosis (cancer)
* Unbalanced cardiovascular pathologies (uncontrolled high blood pressure, coronary artery disease, heart failure, cardiac arrhythmia due to atrial fibrillation)
* Endocrine pathology (hypothyroidism, hyperthyroidism, type 1 diabetes)
* Breathing failure
* Recent hospitalisation (< 30 days)
* Declaration of unstable psychiatric condition (psychosis, depression, bipolar, disorder)
* Chronic medication that may interfere with memory measures or that may alter the quantitative and qualitative parameters of sleep (antidepressants, neuroleptic, antiparkinsonian drugs, corticosteroids, antiepileptics, central analgesics and muscle relaxants)
* Presenting drug and/or alcohol addiction, coffee abuse
* Having an extreme Chronotype (score on Horne and Ostberg Circadian Typology Questionnaire ≤ 30 or ≥ 70)
* Having a moderate or high level of physical activity (categorial score in the International Physical Activity Questionnaire (IPAQ) short version)

Ages: 60 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-01-25 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Change in sleep onset latency measured by polysomnography | Polysomnography is recorded one night before the intervention (baseline) and one night after the intervention (from 12 to 14 weeks after baseline, depending on the intervention).
  Objective measure of sleep quantity expressed in minutes.
Change in total sleep time measured by polysomnography | Polysomnography is recorded one night before the intervention (baseline) and one night after the intervention (from 12 to 14 weeks after baseline, depending on the intervention).
  Objective measure of sleep quantity expressed in minutes.
Change in wake time after sleep onset measured by polysomnography | Polysomnography is recorded one night before the intervention (baseline) and one night after the intervention (from 12 to 14 weeks after baseline, depending on the intervention).
  Objective measure of sleep quantity expressed in minutes.
Change in number of awakenings measured by polysomnography | Polysomnography is recorded one night before the intervention (baseline) and one night after the intervention (from 12 to 14 weeks after baseline, depending on the intervention).
  Objective measure of sleep quantity.
Change in sleep efficiency measured by polysomnography | Polysomnography is recorded one night before the intervention (baseline) and one night after the intervention (from 12 to 14 weeks after baseline, depending on the intervention).
  Objective measure of sleep quantity expressed in % and defined as 100 * total sleep time / time in bed.
Change in percentage of time spent in the different stages sleep measured by polysomnography | Polysomnography is recorded one night before the intervention (baseline) and one night after the intervention (from 12 to 14 weeks after baseline, depending on the intervention).
  Objective measure of sleep quantity expressed in % of time spent in stage 1 sleep, stage 2 sleep, stage 3 sleep and in rapid eye movement (REM) sleep.
Change in sleep quality measured by polysomnography | Polysomnography is recorded one night before the intervention (baseline) and one night after the intervention (from 12 to 14 weeks after baseline, depending on the intervention).
  Objective measure of sleep quality. The variable use to determine sleep quality is the sleep fragmentation index (SFI).
  SFI is defined as the total number of awakenings and any sleep stage shift divided by the total sleep time ; and expressed in number of events per hour.
Change in time in bed measured by actigraphy | Actigraphy is recorded continuously during one week before the intervention (baseline) and one week after the intervention (at 12 and / or 14 weeks after baseline, depending on the intervention).
  Objective measure of sleep quantity, expressed in minutes and based on bedtime and wake time.
Change in sleep onset latency measured by actigraphy | Actigraphy is recorded continuously during one week before the intervention (baseline) and one week after the intervention (at 12 and / or 14 weeks after baseline, depending on the intervention).
  Objective measure of sleep quantity expressed in minutes.
Change in total sleep time measured by actigraphy | Actigraphy is recorded continuously during one week before the intervention (baseline) and one week after the intervention (at 12 and / or 14 weeks after baseline, depending on the intervention).
  Objective measure of sleep quantity expressed in minutes.
Change in wake time after sleep onset measured by actigraphy | Actigraphy is recorded continuously during one week before the intervention (baseline) and one week after the intervention (at 12 and / or 14 weeks after baseline, depending on the intervention).
  Objective measure of sleep quantity expressed in minutes.
Change in sleep efficiency measured by actigraphy | Actigraphy is recorded continuously during one week before the intervention (baseline) and one week after the intervention (at 12 and / or 14 weeks after baseline, depending on the intervention).
  Objective measure of sleep quantity expressed in % and defined as 100 * total sleep time / time in bed.
Change in sleep quality measured by actigraphy | Actigraphy is recorded continuously during one week before the intervention (baseline) and one week after the intervention (at 12 and / or 14 weeks after baseline, depending on the intervention).
  Objective measure of sleep quality. Actigraphic measure of sleep quality is the fragmentation index defined as the sum of the Mobile time (%) and the Immobile bouts <=1min (%).

SECONDARY OUTCOMES:
Change in quality of life | Before the intervention (= baseline) and after the intervention (from 12 to 14 weeks after baseline, depending on the intervention)
  The French version of the SF-36 health survey (Leplège, 2001) includes 11 questions with 5-point rating scales.
  This survey measures eight scales: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, and mental health. For each scale, a score from 0 to 100 is calculated : a higher score means a better quality of live.
  Moreover, from these eight scales, two distinct concepts are measured by the SF-36:
  * a physical dimension, represented by the Physical Component Summary (PCS), and
  * a mental dimension, represented by the Mental Component Summary (MCS)
Change in state anxiety | Before the intervention (= baseline) and after the intervention (from 12 to 14 weeks after baseline, depending on the intervention)
  Part A of the State-Trait Anxiety Inventory (STAI-A ; Spielberger et al., 1970).
  It consists in 20 statements for which volunteers have to evaluate how they feel at a particular moment in time.
  Each answer is scored from 1 to 4, with 1 = low degree of anxiety, and 4 = high degree of anxiety.
  Global score varies from 20 to 80, and means :
  * from 20 to 35 : very low state anxiety
  * from 36 to 45 : low state anxiety
  * from 46 to 55 : medium state anxiety
  * from 56 to 65 : high state anxiety
  * from 66 to 80 : very high state anxiety
Change in visual analog scale of anxiety | Before the intervention (= baseline) and after the intervention (from 12 to 14 weeks after baseline, depending on the intervention)
  Volunteers are asked to place a vertical mark on a 100-mm horizontal line, between "calm" (on the left edge) and "anxious" (on the right edge) (Abend et al., 2014).
Change in the Geriatric Depression Scale | Before the intervention (= baseline) and after the intervention (from 12 to 14 weeks after baseline, depending on the intervention)
  The Geriatric Depression Scale has been designed to specifically rate depression in older adults (Lach et al., 2010; Yesavage et al., 1982).
  This scale includes 30 "yes / no" questions.
  Global score varies between 0 and 30, and means :
  * from 0 to 9 : no depression
  * from 10 to 20 : minor depression
  * from 21 to 30 : major depression
Change in cognitive functions: Stroop test | Before the intervention (= baseline) and after the intervention (from 12 to 14 weeks after baseline, depending on the intervention)
  Evaluation of selective attention. Stroop test has three parts:
  1. - Denomination condition: Volunteers have to name, as fast as possible, the color of rectangles printed in the card A.
  2. - Reading condition: Volunteers have to read, as fast as possible, words printed in black and white in the card B.
  3. - Interference condition: Volunteers have to name, as fast as possible, the color of the words printed in colors in the card C.
  Dependant variables recorded in each condition:
  * Time to perform the task
  * Number of errors = number of self-corrected errors + non-self-corrected errors
  Calculation of interference scores:
  * Time in the Denomination condition - Time in the Interference condition
  * Number of errors in the Denomination condition - Number of errors in the Interference condition
Change in cognitive functions: trail making test (TMT) | Before the intervention (= baseline) and after the intervention (from 12 to 14 weeks after baseline, depending on the intervention)
  Two parts:
  1. TMT-A: Processing speed: volunteers have to link, as fast as possible, numbers from 1 to 25 in sequential order.
  2. TMT-B: Flexibility : volunteers have to alternate, as fast as possible, between numbers from 1 to 13 and letters from A to L : 1-A-2-B-3-C, etc.
  Dependant variables recorded in each part:
  * Time to perform the task
  * Number of errors for TMT-A = number of self-corrected errors + non-self-corrected errors
  * Number of errors for TMT-B = number of self-corrected errors + non-self-corrected errors + perseverative errors
  Scoring procedure:
  * Time to perform TMT-B - Time to perform TMT-A
  * Number of errors for TMT-B - Number of errors for TMT-A
Change in cognitive functions: dual-task Baddeley | Before the intervention (= baseline) and after the intervention (from 12 to 14 weeks after baseline, depending on the intervention)
  Assessment of working memory. First: determination of memory span. Single task 1: memory span for 2 minutes Single task 2: visuo spatial tracking task for 2 minutes Dual-task: both tasks are completed simultaneously for 2 minutes
  Dependant variables recorded:
  * Single task 1: number of correctly recalled series of items
  * Single task 2: number of ticked boxes
  Scoring procedure:
  * Recall performance = (number of correctly recalled series of items during single task - number of correctly recalled series of items during dual-task) / number of correctly recalled series of items during single task.
  * Tracking performance = (number of ticked boxes during single task - number of ticked boxes during dual task) / number of ticked boxes during single task.
  * Mu index (index reflecting the performance decrement due to the dual-task) = (1-((Recall performance + Tracking performance)/2))*100. A high Mu index means high dual-task performance.
Change in long term memory | Before the intervention (= baseline) and after the intervention (from 12 to 14 weeks after baseline, depending on the intervention)
  Computerized memory task, based on the Memory game (Rasch et al., 2007) comprising 24 cards (12 pairs of similar cards).
  Learning condition: Volunteers have to find pairs of identical cards. Learning is completed when volunteers reach at least 68% of correct answers, i.e. when 16 cards are correctly assembled on 24.
  Recall condition takes place the next morning. Only one trial is performed.
  Dependant variables recorded:
  * Number of pairs correctly recalled during the learning condition
  * Number of pairs correctly recalled the next morning
  Scoring procedure:
  - Delta index: (number of pairs correctly recalled the next morning - number of pairs correctly recalled during the learning condition) / number of pairs correctly recalled during the learning condition
Change in Hand grip strength | Before the intervention (= baseline) and after the intervention (from 12 to 14 weeks after baseline, depending on the intervention)
  The hand grip strength is measured with a dynamometer. Volunteers complete three trials per hand, during 3 to 5 secondes, with 1-minute break between each trial to minimize fatigue effects.
  Among the six measures, maximum values of each hand are retained (expressed in kg).
Change in Leg extension power | Before the intervention (= baseline) and after the intervention (from 12 to 14 weeks after baseline, depending on the intervention)
  Leg extension power is assessed with the Nottingham power rig. Seated volunteers have to extend their tested leg (right leg) as fast and hard as possible by pushing unilaterally the footplate. There are eight trials, with 30-second break in between.
  Dependant variables recorded:
  * maximal leg power (expressed in watts)
  * maximal leg power relative to the weight of the individual (expressed in watts/kg)
Change in Postural balance | Before the intervention (= baseline) and after the intervention (from 12 to 14 weeks after baseline, depending on the intervention)
  Postural balance is assessed through the Synapsys posturography system (Synapsys Inc.).
  Volunteers stand on the Synapsys posturography system, feet apart, with their arms alongside their body, looking straight ahead.
  Postural balance is measured in two conditions, with eyes open and eyes closed. There are two 30-second trials per condition.
  For each trial, the position of the center of pressure (CoP) is recorded. Limit of stability test is recorded without time limitation. The maximum amplitude of oscillations of the CoP in mediolateral and anterioposterior directions are recorded.
Change in maximum incremental cardiopulmonary test | Before the intervention (= baseline) and after the intervention (from 12 to 14 weeks after baseline, depending on the intervention)
  The maximum incremental cardiopulmonary test is performed on an ergometric bicycle, based on an individualized protocol.
  Prior to the test, a resting ECG is performed and verified by a cardiologist. Following a 3 min warm-up (30 watts), the power is incremented by 20 watts every 2 minutes until exhaustion. The test is followed by a 3-minute recovery period.
  Maximum effort is determined by the occurrence of the following two criteria:
  * 1) Presence of a VO2 plateau despite an increase of power (Åstrand et al., 1994);
  * 2) Increase in oxygen consumption of the last increment should not exceed 100 ml/min despite the increase in power (Di Prampero et al., 1993).
  Dependant variables recorded:
  * Maximum oxygen consumption (VO2 max)
  * Maximum aerobic power
  * Maximum heart rate
  * Respiratory quotient (RQ) at the end of test (RQ = Volume of CO2 / Volume of O2)
Change in the Global Physical Activity Questionnaire (GPAQ) | Before the intervention (= baseline) and after the intervention (from 12 to 14 weeks after baseline, depending on the intervention)
  Questionnaire developed by the World Health Organization, which consists in 19 questions grouped to capture physical activity undertaken in different behavioural domains, as work, transport and discretionary (also known as leisure or recreation) (Cleland and al., 2014).
  Within the work and discretionary domains, questions assess the frequency and duration of two different categories of activity defined by the energy requirement or intensity (vigorous or moderate intensity).
  In the transport domain, the frequency and duration of all walking and cycling for transport is captured but no attempt is made to differentiate between these activities.
  One additional item collects time spent in sedentary activities.
  Calculation of a global MET score (Metabolic Equivalent of Task, 1 MET = 1 kcal/kg/hour).
  Higher MET score means high physical activity.
Change in Timed up and go test | Before the intervention (= baseline) and after the intervention (from 12 to 14 weeks after baseline, depending on the intervention)
  Assessment of dynamic balance in the older adults (Mathias et al., 1986; Podsiadlo & Richardson, 1991).
  Volunteers are asked to sit down on a chair with their feet on the floor and their hands on their legs. At the "go" signal, they have to stand up, walk 3 meters, turn around a cone, walk back, and sit down again.
  The performance time starts when volunteers start moving to stand up and ends when they sit down again properly.
  The test is performed in two conditions:
  * Two trials at a self-paced velocity, and
  * Two trials as fast as possible
  Duration of the two best trials of the two conditions are retained (Podsiadlo & Richardson, 1991).

CONTACTS AND LOCATIONS:
Overall Officials: Hervé Hervé, M.D. PhD., Principal Investigator — Université de Caen Normandie, U1075 COMETE Inserm
Locations (1):
- Antoine Langeard, Caen, France